CLINICAL TRIAL: NCT03569527
Title: Kiwifruit, Prunes, & Fiber for Abdominal and Bowel Symptoms in US Patients With Chronic Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Shanti Eswaran, Clinical Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00127778
Record Dates: First submitted 2018-06-11; First posted 2018-06-26 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Chronic Constipation
Keywords: Kiwifruit
MeSH Terms: interventions — alcohol acyltransferase, Actinidia; Dietary Fiber

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kiwifruit (Active Comparator): Treating chronic constipation with 2 kiwifruit (6g fiber) per day
  Interventions: Dietary Supplement: Kiwifruit
- Psyllium fiber (Active Comparator): Treating chronic constipation with 24g psyllium fiber (6g fiber) per day
  Interventions: Dietary Supplement: Fiber
- Prune (Active Comparator): Treating chronic constipation with 100g dried plums (6g fiber) per day
  Interventions: Dietary Supplement: Prunes

INTERVENTIONS:
Dietary Supplement: Kiwifruit — The total duration of the study will be 8 weeks (2- week baseline, 4-week intervention, and 2-week follow-up). Eligible patients will be randomized to receive kiwifruit (2 green kiwifruit per day for the 4 week intervention period.
  Arms: Kiwifruit
Dietary Supplement: Fiber — The total duration of the study will be 8 weeks (2- week baseline, 4-week intervention, and 2-week follow-up). Eligible patients will be randomized to receive psyllium fiber (24 g/day, fiber=6g/day) for the 4 week intervention period.
  Arms: Psyllium fiber
Dietary Supplement: Prunes — The total duration of the study will be 8 weeks (2- week baseline, 4-week intervention, and 2-week follow-up). Eligible patients will be randomized to receive prunes/dried plums (100g, fiber=6 g/day) for the 4 week intervention period.
  Other Names: Dried Plums
  Arms: Prune

SUMMARY:
This is a parallel group pilot study comparing the efficacy green kiwifruit, prunes or psyllium on abdominal and bowel related symptoms in US patients with chronic constipation patients.

DETAILED DESCRIPTION:
Chronic constipation and Irritable Bowel Syndrome with constipation are common gastrointestinal disorders which negatively impact quality of life, reduce work productivity, and account for significant direct and indirect costs. Patients with CC and IBS-C suffer with bowel symptoms such as reduced stool frequency, hard stool consistency, straining or a sensation of incomplete evacuation. Coupled with barriers which limit access to expensive prescription increasing concerns regarding the long-term safety of chronically dosed medications and, there has been an increasing demand for more "natural" solutions to a wide range of medical conditions, including CC and IBS-C. Green kiwifruit has long been used as a natural remedy to improve GI complaints. A growing body of literature supports the benefits of kiwifruit for gut health and in particular, abdominal discomfort and bowel regularity. In addition, patients are interested in dietary changes that could improve their symptoms The investigators propose a parallel group pilot study comparing the efficacy green kiwifruit, prunes or psyllium on abdominal and bowel related symptoms in US patients with chronic constipation patients. The investigators plan to recruit chronic constipation patients with or without pain. The total duration of the study will be 8 weeks (2- week baseline, 4-week intervention, and 2-week follow-up). Eligible patients will be randomized to receive kiwifruit (2 green kiwifruit per day, psyllium (12 g b.d./day, fiber=6g/day) or dried plums (50 g b.d., fiber=6 gm/day) for the 4 week intervention period. It is expected that Kiwifruit will offer greater efficacy than psyllium and prunes for abdominal and bowel symptoms in US patients with chronic constipation. This will be the first US data addressing the efficacy of Kiwifruit for abdominal and bowel symptoms in patients with chronic constipation.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of functional constipation according to modified ROME IV diagnostic criteria*5b i. Must include two or more of the following:

1. Straining more than 25% of defecations
2. Lumpy or hard stools more than 25% of defecations
3. Sensation of incomplete evacuation more than 25% of defecations
4. Sensation of anorectal obstruction/blockage more than 25% of defecations
5. Manual manoeuvres to facilitate more than 25% of defecations (e.g. digital evacuation, support of pelvic floor)
6. Fewer than three defecations per week ii. Loose stools are rarely present without the use of laxatives * Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis For the purposes of this study, patients with abdominal pain will be included, but patients with severe pain (defined as average daily abdominal pain score of 7 or higher during the screening period) will be excluded. Patients with an appropriate level of GI symptoms despite taking stable doses (>3 months) of SSRI's, tricyclics or SNRIs will be allowed to enroll.

Exclusion Criteria:

Potential participants will be excluded if they have alarm features (GI bleeding, weight loss, unexplained iron deficiency anaemia, significant family history of colorectal cancer or IBD), anal fissures, significant chronic diseases (cardiovascular, cancer, renal failure, inflammatory bowel disease), previous gastrointestinal surgery (except appendectomy or cholecystectomy), neurological diseases (e.g. multiple sclerosis, spinal cord injury, CVA).

Patients taking opiates will not be eligible to participate. Women who are pregnant, breastfeeding or planning a pregnancy in the 2 months post selection (trial period) will be excluded.

As above, patients with severe IBS symptoms will be excluded (defined as average daily abdominal pain score of 7 or higher during the screening period).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
: Change in complete spontaneous bowel movement (CSBM) | 8 weeks
  Complete spontaneous bowel movement will be recorded. This will be compared to the baseline, run-in periods, and follow-up period.

SECONDARY OUTCOMES:
Change in SBM (spontaneous bowel movements) | 8 weeks
  Spontaneous bowel movements will be recorded. This will be compared to the baseline, run-in periods, and follow-up period.
stool consistency | 8 weeks
  Bristol stool form scale (1-7, lower scores are consistent with constipation; higher scores are consistent with diarrhea) will be recorded. This will be averaged and compared to the baseline, run-in period, and follow-up period.
straining | 8 weeks
  5 point Likert scale for straining will be recorded (1-5, lower scores= less straining, higher scores = more straining). This will be averaged and compared to the baseline, run-in periods, and follow-up period.
abdominal pain | 8 weeks
  Daily score (0-10) for abdominal pain will be recorded (0=no pain, 10= severe pain). This will be averaged and compared to the baseline, run-in periods, and follow-up period.
abdominal discomfort | 8 weeks
  Daily score (0-10) for abdominal discomfort will be recorded (0=no pain, 10= severe pain). This will be averaged and compared to the baseline, run-in periods, and follow-up period.
bloating | 8 weeks
  Daily score (0-10) for abdominal bloating will be recorded (0=no pain, 10= severe pain). This will be averaged and compared to the baseline, run-in periods, and follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Shanti Eswaran, MD, Principal Investigator — Department of Internal Medicine, Division of Gastroenterology, University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chey SW, Chey WD, Jackson K, Eswaran S. Exploratory Comparative Effectiveness Trial of Green Kiwifruit, Psyllium, or Prunes in US Patients With Chronic Constipation. Am J Gastroenterol. 2021 Jun 1;116(6):1304-1312. doi: 10.14309/ajg.0000000000001149. PMID 34074830
- [Derived] Dimidi E, Staudacher HM. Could a kiwifruit a day keep the doctor away? Lancet Gastroenterol Hepatol. 2020 Jul;5(7):648. doi: 10.1016/S2468-1253(20)30163-1. No abstract available. PMID 32553145